CLINICAL TRIAL: NCT06586931
Title: Accuracy of Venous Excess Ultrasound (VEXUS) Score Versus Central Venous Pressure to Assess Volume Status in Patients With Severe Sepsis
Brief Title: Accuracy of Venous Excess Ultrasound (VEXUS) Score Versus Central Venous Pressure in Patients With Severe Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Andrew Emad Thabet Ebrahim, Accuracy of venous excess ultrasound (VEXUS) score versus central venous pressure to assess volume status in patients with severe sepsis, Minia University
Other Study IDs: VEXUS score in severe sepsis
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sepsis, Severe
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assessing septic patients with a noninvasive ultrasound protocol, and earlier identification of fluid overload to help clinicians decide whether to administer supplemental fluid therapy or suspend its administration and to evaluate the possible relation between the different VExUS grades and the adverse effects of intensive fluid administration

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction caused by a poorly regulated host response to infection. Septic shock is still a leading cause of death worldwide as it can induce multi-organ failure (1).

Septic shock is a subset of sepsis with manifest circulatory dysfunction .intravenous fluid therapy is an essential intervention to promote hemodynamic stabilization.. Similarly, septic patients are a very different and difficult subset in intensive care unit (ICU). They are vasodilated and require fluid resuscitation for optimization of venous volume and cardiac output (2).

Central venous pressure measurement which has been used for ages, is not the ideal monitoring technique as it does not correlate with blood volume and does not give a true representation of the response of fluid challenge (3).

a venous excess Doppler ultrasound (VExUS) grading system, are parameters for the assessment of the fluid status of the patient and organ congestion. This protocol evaluates the amount of venous congestion in the abdominal organs, specifically by scanning the portal, hepatic, and intrarenal veins. Doppler interrogation of these vessels yields a specific pattern corresponding to a level of venous congestion: normal, mild, or severe. (4).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years old) with the diagnosis of severe sepsis and clinical indication to be admitted in critical care units are recruited. Sepsis should be suspected to be the primary cause of their acute illness by the treating physician, consistent with the

Surviving Sepsis Campaign Guidelines (2021) :

* Life-threatening organ dysfunction
* Diagnosis of infection Some patients diagnosed with sepsis will not meet the criteria, but will be eligible for the study if the treating physician makes a clinical diagnosis of severe sepsis.

Exclusion Criteria:

* 1. Refusal to participate 2. Patients in hemodialysis program 3. Patients with previously known conditions that interfere with portal Doppler assessments, namely liver cirrhosis, or severe tricuspid regurgitation with structural heart disease. If any of these conditions are identified during the present episode, the patient would also be excluded.

  4. Age < 18 years 5. Patients subjected to withdrawal of care 6. Hemodynamic instability due to active hemorrhage 7. Acute coronary syndrome 8. Indication for immediate surgery 9. Received CPR within 24 hours of enrollment 10. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (≥ 18 years old) with the diagnosis of severe sepsis and clinical indication to be admitted in critical care units are recruited. Sepsis should be suspected to be the primary cause of their acute illness by the treating physician,
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
VEXUS score | Baseline
  Assessment of fluid status in septic patients by VEXUS score

SECONDARY OUTCOMES:
Accuracy of CVP for assessment of fluid status in septic patients | Baseline
  Comparison of CVP with VEXUS score to assess fluid status

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Zekry, Professor, Study Chair — Minia U

REFERENCES:
- [Background] Longino A, Martin K, Leyba K, Siegel G, Gill E, Douglas IS, Burke J. Correlation between the VExUS score and right atrial pressure: a pilot prospective observational study. Crit Care. 2023 May 26;27(1):205. doi: 10.1186/s13054-023-04471-0. PMID 37237315
- [Background] Rola P, Miralles-Aguiar F, Argaiz E, Beaubien-Souligny W, Haycock K, Karimov T, Dinh VA, Spiegel R. Clinical applications of the venous excess ultrasound (VExUS) score: conceptual review and case series. Ultrasound J. 2021 Jun 19;13(1):32. doi: 10.1186/s13089-021-00232-8. PMID 34146184
- See also: VEXUS score verses central venous pressure — http://pubmed.ncbi.nlm.nih.gov/37237315/